CLINICAL TRIAL: NCT05747417
Title: Prismatic Correction for Improving Near Visual Acuity in Patients With Maculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Shifa Trust Eye Hospital (Other)
Responsible Party: Principal Investigator, Mehreen Tanveer, Manager Light House, Al-Shifa Trust Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AlShifaTrust Eye
Record Dates: First submitted 2023-01-25; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prism glasses (Experimental): prisms glasses are advised with ranging of 4prism diopters to 10 prism diopters
  Interventions: Other: prismatic glasses
- presbyopic glasses (No Intervention): simple presbyopia glasses according to age are advised

INTERVENTIONS:
Other: prismatic glasses — prism glasses ranging from 4-10 prism diopters
  Arms: prism glasses

SUMMARY:
patients with maculopathy reported in low vision clinic are tested for prismatic glasses for near vision. The pre and post visual acuity was recorded.

DETAILED DESCRIPTION:
Diagnosed patient of maculopathy who was visited in low vision clinic are divided in two groups , one is control group (prescribed simple near vision glasses) and other is interventional group(prescribed prismatic glasses). Both groups were follow up after one month to check the improvement in near visual acuity

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed patients of maculopathy refer to low vision clinic
2. Patients with both genders
3. VA from LogMAR 1.0 to LogMAR 0.3

Exclusion Criteria:

1. Maculopathy patients with other ocular disease
2. VA worsen the LogMAR 1.0
3. Patients with mental illness and other physical lmitations

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Prismatic Correction for Improving Near Visual Acuity in Patients with Maculopathy | 7 -8 months
  A Per forma/questionnaire is used to document Near visual Acuity with the help of light house Chart to see improvement in visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Al Shifa Trust Eye Hospital Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No